CLINICAL TRIAL: NCT00954460
Title: Multicenter Open-Label Treatment Protocol to Observe the Safety of Gene-Activated™ Human Glucocerebrosidase (GA-GCB, Velaglucerase Alfa) ERT in Newly Diagnosed or Previously Treated (With Imiglucerase) Patients With Type 1 Gaucher Disease
Brief Title: Treatment Protocol of Velaglucerase Alfa for Patients With Type 1 Gaucher Disease
Status: Approved for marketing | Type: Expanded Access
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: HGT-GCB-058
Record Dates: First submitted 2009-08-05; First posted 2009-08-07 (Estimated); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Gaucher Disease, Type 1
Keywords: VPRIV; Enzyme Replacement Therapy; Gaucher disease; glucocerebrosidase; beta-glucocerebrosidase; Acid beta-glucocerebrosidase; glucosylceramidase; D-glucosyl-N-acylsphingosine glucohydrolase; gene activation; human
MeSH Terms: conditions — Gaucher Disease | interventions — Glucosylceramidase

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: velaglucerase alfa — up to 60 U/kg, every other week via intravenous infusion
  Other Names: VPRIV; Gene activated human glucocerebrosidase; GA-GCB

SUMMARY:
Gaucher disease is a rare lysosomal storage disorder caused by the deficiency of the enzyme glucocerebrosidase (GCB). Due to the deficiency of functional GCB, glucocerebroside accumulates within macrophages leading to cellular engorgement, organomegaly, and organ system dysfunction. The purpose of this treatment protocol is to observe the safety of velaglucerase alfa in patients with type 1 Gaucher disease who are either treatment naive (newly diagnosed) or who are currently being treated with the Enzyme Replacement Therapy (ERT) imiglucerase.

DETAILED DESCRIPTION:
Type 1 Gaucher disease, the most common form, accounts for more than 90% of all cases of Gaucher disease and does not involve the CNS. Typical manifestations of type 1 Gaucher disease include hepatomegaly, splenomegaly, thrombocytopenia, bleeding tendencies, anemia, hypermetabolism, skeletal pathology, growth retardation, pulmonary disease, and decreased quality of life. Velaglucerase alfa (Gene-Activated™ human glucocerebrosidase;GA-GCB) is produced in a continuous human cell line using proprietary gene-activation technology and has an identical amino acid sequence to the naturally occurring human enzyme. Velaglucerase alfa contains terminal mannose residues that target the enzyme to the macrophages-the primary target cells in Gaucher disease. This treatment protocol will observe the safety of velaglucerase alfa in patients with type 1 Gaucher disease who are either treatment naive (newly diagnosed) or who are currently being treated with the Enzyme Replacement Therapy (ERT) imiglucerase. Patients currently being treated with ERT for their Gaucher disease will receive the same number of units of velaglucerase alfa per month as their imiglucerase dose for doses between 30-120 U/kg/month. For patients who experienced dose reductions in their imiglucerase treatment due to supply constraints the pre-reduction monthly dose may be used to determine the monthly dose of velaglucerase alfa.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has a documented diagnosis of type 1 Gaucher disease
2. The patient is > 2 years of age
3. The patient has NOT previously experienced an anaphylactic or anaphylactoid reaction to another ERT including imiglucerase
4. Women of child-bearing potential must agree to use a medically acceptable method of contraception at all times during the study; and must have a negative result to a pregnancy test as required throughout their participation in the study. Male patients must use a medically acceptable method of birth control throughout their participation in the study and must report their partner's pregnancy.
5. The patient is sufficiently cooperative to participate in this treatment plan as judged by the Investigator
6. If the patient is naïve or new to treatment, the patient has one or more of the following (in absence of the following criteria, please call the sponsor for treatment justification):

   * Gaucher disease-related anemia
   * Moderate splenomegaly (2 to 3 cm below the left costal margin), by palpation
   * Gaucher disease-related thrombocytopenia
   * Gaucher disease-related palpable enlarged liver

Exclusion Criteria: None

Min Age: 3 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (32):
- United States (32):
  - St Joseph's Hospital & Medical Center, Phoenix, Arizona
  - Tower Hematology Oncology, Beverly Hills, California
  - Rady's Children's Hospital of San Diego, La Jolla, California
  - Southern California Permanente Medical Group, Los Angeles, California
  - The Permanente Medical Group, Sacramento, California
  - Stanford University Medical Genetics, Stanford, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - University Research Foundation for Lysosomal Storage Diseases, Coral Springs, Florida
  - Gainesville Hematology Oncology Associates, Gainesville, Florida
  - Adventis Healthcare System dba Florida Hospital, Orlando, Florida
  - East Lake Oncology, Palm Harbor, Florida
  - Emory Genetics, Decatur, Georgia
  - Children's Memorial Hospital, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Annapolis Oncology Center, Annapolis, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - University of Massachusetts, Shrewsbury, Massachusetts
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - The University Research Foundation for Lysosomal Storage Diseases, Kansas City, Missouri
  - St. Joseph's, Paterson, New Jersey
  - Hemophilia Center of Western New York Incorporated, Buffalo, New York
  - North Shore Hematology/Oncology - Manhasset, Manhasset, New York
  - New York University School of Medicine, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Fullerton Genetic, Asheville, North Carolina
  - Duke Medical Center, Durham, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Virginia Health Systems, Charlottesville, Virginia
  - O & O Alpan, LLC, Springfield, Virginia

REFERENCES:
- [Derived] Pastores GM, Rosenbloom B, Weinreb N, Goker-Alpan O, Grabowski G, Cohn GM, Zahrieh D. A multicenter open-label treatment protocol (HGT-GCB-058) of velaglucerase alfa enzyme replacement therapy in patients with Gaucher disease type 1: safety and tolerability. Genet Med. 2014 May;16(5):359-66. doi: 10.1038/gim.2013.154. Epub 2013 Nov 21. PMID 24263462